CLINICAL TRIAL: NCT06950268
Title: A Randomized Controlled Trial Comparing Active and Passive Motion Splint Immobilization for the Treatment of Extensor Tendon Injuries in Zones IV to VI of the Hand
Brief Title: Randomized Trial of Active vs Passive Splinting for Extensor Tendon Injuries in Zones IV to VI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/307
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hand Injuries; Tendon Injuries
Keywords: Classic Immobilization; Hand Surgery; Postoperative Rehabilitation; Extensor Tendon Repair; ICAMS; Finger Tendon; Zones IV to VI; Controlled Motion Splint
MeSH Terms: conditions — Hand Injuries; Tendon Injuries | interventions — Splints

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, parallel-group design comparing ICAMS versus classic immobilization following extensor tendon tenorrhaphy
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind study. The outcomes assessor was blinded to group allocation. Participants and care providers were not blinded due to the visible nature of the splints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICAMS Group (Experimental): Participants received immediate controlled active motion splinting (ICAMS) after extensor tendon tenorrhaphy. The ICAMS protocol included a daytime yoke splint, which maintained the injured finger in 20° more extension than adjacent fingers, and a nocturnal intrinsic plus static splint. The protocol was maintained for 4 weeks post-surgery
  Interventions: Device: ICAMS Splinting Protocol
- Classic Immobilization Group (Active Comparator): Participants received standard immobilization with a plaster splint in the intrinsic plus position following extensor tendon tenorrhaphy. The immobilization was maintained continuously for 4 weeks.
  Interventions: Device: Classic Plaster Immobilization

INTERVENTIONS:
Device: ICAMS Splinting Protocol — The ICAMS protocol consisted of a daytime yoke splint maintaining the injured finger in 20° more extension than adjacent fingers, combined with a nocturnal static splint in the intrinsic plus position. The splinting was applied for 4 weeks following extensor tendon tenorrhaphy.
  Other Names: Immediate Controlled Active Motion Splinting; Dynamic Splint; Yoke Splint
  Arms: ICAMS Group
Device: Classic Plaster Immobilization — Participants received a classic plaster splint in the intrinsic plus position worn continuously for 4 weeks following extensor tendon tenorrhaphy.
  Other Names: Intrinsic Plus Position Splint; Standard Immobilization
  Arms: Classic Immobilization Group

SUMMARY:
This study compares two methods of post-operative immobilization after surgical repair (tenorrhaphy) of extensor tendons in the fingers. Patients were randomly assigned to receive either a standard plaster splint or an alternative splinting method that allows controlled finger movement (ICAMS). The main goal was to determine which method leads to better recovery in terms of finger mobility, grip strength, pain, and patient comfort.

DETAILED DESCRIPTION:
Extensor tendon injuries of the hand are commonly treated with immobilization for 4-6 weeks using a plaster splint in the intrinsic plus position. However, prolonged immobilization may lead to tendon adhesions, joint stiffness, and delayed return to function. This randomized controlled clinical trial evaluated the efficacy of an immediate controlled active motion splinting protocol (ICAMS) compared to classic immobilization (CI) following extensor tendon tenorrhaphy in zones IV, V, and VI. Thirty patients were randomly assigned to either group. Functional outcomes were assessed at 4 and 6 weeks post-injury, including grip strength, joint range of motion, pain (VAS), Quick-DASH score, and patient satisfaction. The ICAMS group showed significantly better results in all main functional parameters. These findings support the use of early active motion protocols in selected cases of extensor tendon injury to enhance recovery and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Patients from the CHUVI Health Area
* Diagnosed with an acute, single, complete extensor tendon laceration in zones IV, V, or VI of the long fingers
* Treated with primary tenorrhaphy
* Provided signed informed consent
* Agreed to attend follow-up visits and comply with the study protocol

Exclusion Criteria:

* More than one extensor tendon laceration in the same hand
* Injuries involving the thumb
* Tendon injuries with loss of substance
* Associated injuries at the same level (e.g., bone fracture, nerve lesion)
* Patients with cognitive impairment or inability to follow the protocol
* Presence of other injuries or medical conditions that could interfere with assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Grip Strength of the Injured Hand | 4 and 6 weeks after injury
  Grip strength was measured using a JAMAR manual dynamometer to evaluate functional recovery after extensor tendon tenorrhaphy. Measurements were taken at 4 and 6 weeks post-injury.

SECONDARY OUTCOMES:
Change in MCP Joint Flexion | 4 and 6 weeks after injury
  Active flexion of the metacarpophalangeal (MCP) joints of the injured finger was measured to assess recovery of joint mobility.
Pain Intensity (VAS Score) | 4 and 6 weeks after injury
  Pain was evaluated using a 10-point Visual Analog Scale (VAS) at both follow-up visits.
Quick-DASH Score | 4 and 6 weeks after injury
  Upper limb disability and function were assessed using the Quick Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) questionnaire.
Patient Comfort With Immobilization | 4 and 6 weeks after injury
  Patients rated their comfort with the splint using a yes/no response at 4 weeks post-treatment.
Patient Satisfaction With Treatment Outcome | 4 and 6 weeks after injury
  Patients reported overall satisfaction with the treatment using a yes/no response.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Cela-López, MD, Principal Investigator — Sergas
Locations (1):
- CHUVI Hospital (Complejo Hospitalario Universitario de Vigo), Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No